CLINICAL TRIAL: NCT00917787
Title: Analysis of Blood-based Biomarkers of Asthma
Acronym: ABBA
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: H6788-34128-01
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — sputum, saliva, DNA, RNA, Plasma, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy, Non-asthmatic
- Asthma

SUMMARY:
The purpose of this study is to analyze markers of inflammation in blood and in induced sputum for the purpose of identifying molecular markers of specific asthma phenotypes. The investigators' specific interest is demonstrating that periostin levels are higher than normal in blood. The investigators already have solid preliminary data to support this hypothesis, and our goal here is to replicate preliminary findings and extend them by examining further the characteristics of the asthma subgroup with elevated periostin levels.

DETAILED DESCRIPTION:
This is a cross-sectional study in patients with asthma and healthy controls in which we will analyze markers of inflammation in blood and in induced sputum for the purpose of identifying molecular markers of specific asthma phenotypes. Our specific interest in demonstrating that periostin levels are higher than normal in blood. We already have solid preliminary data to support this hypothesis, and our goal here is to replicate preliminary findings and extend them by examining further the characteristics of the asthma subgroup with elevated periostin levels. In this regard, we propose detailed phenotyping of the asthmatic subjects and the healthy controls, including measures in induced sputum, exhaled air and detailed physiologic measures including measures of airflow, lung volumes, and methacholine responsiveness. In earlier work we have found that periostin is a marker of Th-2 driven asthma, and we will use the data collected here to further explore this possibility. The biospecimens collected here will also allow us to expand existing plasma, DNA, RNA, and sputum samples in the UCSF Airway tissue bank, so that we can continue to build this resource for future research questions.

ELIGIBILITY:
Asthmatic Subjects Inclusion criteria

1. Male and female subjects between the ages of 18 and 70 years with a history of asthma who may or may not be taking inhaled corticosteroids for asthma control.
2. Physician diagnosis of asthma
3. PC20FEV1 methacholine ≤ 8.0 mg/mL, except for those taking daily inhaled corticosteroids, for which the PC20 methacholine should be < 16 mg/mL.
4. Ability to provide informed consent.

Healthy Subjects Inclusion criteria

1. Healthy male and female subjects with no history of asthma between the ages of 18 and 70 years. Subjects should not be taking inhaled or oral corticosteroids.
2. No lifetime history of asthma or allergic rhinitis.
3. Ability to provide informed consent.

Exclusion Criteria for both subject groups

1. Lung disease other than asthma.
2. History of an upper or lower respiratory tract infection in the 4 weeks preceding the study.
3. Females who are pregnant or breast-feeding
4. Subjects must be non-smokers (patients who have never smoked or patients who have smoked ≤5 cigarettes per month and have a total pack-year smoking history < 10 packs).
5. Use of marijuana >1 time per month in the last year and use of marijuana in the 6 weeks prior to enrollment
6. Use of recreational drugs other than marijuana in the 12 months preceding the study.
7. Use of Beta blocker medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asthmatics and Non-asthmatics
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
periostin levels in blood | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States